CLINICAL TRIAL: NCT00576433
Title: An Open Label Study to Evaluate the Safety and Effect on Treatment Response of MabThera in Patients With Rheumatoid Arthritis Following Inadequate Response to One Prior Anti-TNF Inhibitor
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to a Single Anti-TNF Inhibitor.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21271
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Methotrexate; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: Methotrexate — As prescribed
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15

SUMMARY:
This single arm study will evaluate the safety and efficacy of MabThera in patients with active rheumatoid arthritis who are receiving methotrexate treatment, and who have had an inadequate response to one anti-TNF alpha therapy. All patients will receive MabThera 1000mg i.v. on days 1 and 15, in addition to concomitant methotrexate. Patients who achieve a clinically relevant response to the first course of treatment may be eligible to receive one re-treatment course of MabThera between weeks 24 and 48. The anticipated time on study treatment is 3-12 months, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* moderate to severe active rheumatoid arthritis;
* inadequate response to previous or current treatment with 1 anti-TNF agent;
* receiving methotrexate at a dose of 10-25mg/week for 12 weeks prior to start of study, at a stable dose for >=4 weeks.

Exclusion Criteria:

* previous treatment with MabThera;
* use of an anti-TNF alpha agent within 8 weeks of study start;
* concurrent treatment with any DMARD other than methotrexate;
* active infection, or history of serious recurrent or chronic infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
AEs, including infusion-related adverse events | For 48 weeks after initial treatment

SECONDARY OUTCOMES:
Safety of re-treatment (AEs) | For 24 weeks after re-treatment.
Laboratory parameters, vital signs. | Throughout study
ACR 20/50/70, Eular response rates, DAS 28, ACR core components, HAQ, FACIT. | For 48 weeks after initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Russia (17):
  - Chelyabinsk
  - Irkutsk
  - Kazan'
  - Khabarovsk
  - Khanty-Mansiysk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Ryazan
  - Saint Petersburg
  - Tyumen
  - Ufa
  - Vladivostok
  - Voronezh
  - Yaroslavl
  - Yekaterinburg